CLINICAL TRIAL: NCT04418609
Title: Neuro-COVID-19: Neurological Complications of COVID-19
Acronym: Neuro-COVID
Status: Completed | Type: Observational
Sponsor: Emanuela Keller (Other)
Responsible Party: Sponsor-Investigator, Emanuela Keller, Prof. Dr. Emanuela Keller, University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: Neuro-COVID-19
Record Dates: First submitted 2020-05-28; First posted 2020-06-05 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Neurologic Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: further processing of health data — further processing of biological materials and health related personal data for research
  Other Names: further processing of biological materials and health related personal data

SUMMARY:
The prevalence and typical patterns of neurological complications in hospitalized COVID-19 patients admitted to the intensive care units of the University Hospital Zurich will be investigated. The impact of neurological complications among COVID-19 patients on mortality, functional outcome, and organizational outcomes will be analyzed.

DETAILED DESCRIPTION:
This study is a prospective observational cohort study to document prevalence and severity of neurological symptoms among patients requiring critical care admission for confirmed novel coronavirus disease (COVID-19). COVID-19 is classified as severe acute respiratory syndrome 2 (SARS-CoV-2) and shares significant structural and biological similarities with SARS-CoV, which has neuroinvasive properties and brainstem involvement. Early reports of COVID-19 progression indicate presence of severe neurological complications, including seizures, coma, encephalitis, and cerebrovascular events including ischemic stroke, intracranial hemorrhage, and cerebral venous sinus thromboses. In addition, recent data from Zika-virus and H1N1 influenza pandemics reveal a high incidence of neurological complications, including Guillain Barré syndrome and neonatal microcephaly for Zika-virus and narcolepsy with H1N1 infections. Early reports from China suggest neurological symptoms may occur in approximately 36% of SARS-CoV-2 positive patients, with increased prevalence among more severe cases, and fall into three categories: central nervous system symptoms or diseases, peripheral nervous system symptoms, and skeletal muscular symptoms. However, the exact prevalence of these conditions and impact on patient disease severity and outcomes is unknown. As the incidence and severity of COVID-19 infection continues to rapidly rise on an international level, it is imperative to capture prospective data to accurately document prevalence, severity and clinical characterization of neurological components of COVID-19, the influence of treatment regimens of neurological complications, and role of these confounders on patient and organizational outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age > 18 years old) treated at ICUs
* Admitted with confirmed COVID-19 infection
* Patient exhibiting acute neurological manifestations
* General consent of the Institute of Intensive Care Medicine available from patient or legal representative

Exclusion Criteria:

* Pre-existing severe neurologic dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the Intensive Care Units (ICUs) of the Institute of Intensive Care Medicine, University Hospital of Zurich meeting eligibility criteria during the pandemic will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-09 (Actual)

PRIMARY OUTCOMES:
Prevalence of neurological complications | through study completion, on an average of 3 weeks
  Determine the prevalence of neurological complications in hospitalized COVID-19 patients admitted to the intensive care unit.
Prevalence and outcome of severe neurological complications | through study completion, on an average of 3 weeks
  Examine if empiric COVID-19 therapies are associated with difference in the prevalence and outcome of severe neurological complications of COVID-19.
Impact of neurological complications | through study completion, on an average of 3 weeks
  Determine the impact of neurological complications among COVID-19 patients on mortality, functional outcome, and organizational outcomes (ICU length of stay, hospital length of stay) among patients with confirmed COVID-19.
Characteristic patterns in cerebral imaging and electroencephalography (EEG), as well as cerebrospinal fluid (CSF) | through study completion, on an average of 3 weeks
  Analyze characteristic patterns in cerebral imaging and electroencephalography (EEG), as well as cerebrospinal fluid (CSF) of patients, in whom a lumbar puncture has been performed for clinical reasons
Brain for pathological changes and histopathological findings (if patient dies). | through study completion, on an average of 3 weeks
  Analyze the brain for pathological changes and histopathological findings, if the patient dies.

CONTACTS AND LOCATIONS:
Overall Officials: Emanuela Keller, Prof. Dr., Principal Investigator — University Hospital, Zürich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No